CLINICAL TRIAL: NCT07044726
Title: Betadine vs Sterile Water for Periurethral Preparation Prior to Straight Catherization in the Clinic Setting: A Randomized Controlled Trial
Brief Title: Betadine vs Sterile Water for Periurethral Preparation
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Ankita Gupta, Associate Fellowship Director of Urogynecology and Pelvic Reconstructive Surgery, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 25.0260
Record Dates: First submitted 2025-06-16; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Catherization; Urinary Tract Infection Bacterial
Keywords: Betadine; Sterile Water; Catherization
MeSH Terms: interventions — Povidone-Iodine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Betadine (Active Comparator): Betadine periurethral preparation
  Interventions: Drug: Povidone-Iodine
- Sterile Water (Sham Comparator): Sterile Water periurethral preparation
  Interventions: Drug: Sterile water

INTERVENTIONS:
Drug: Povidone-Iodine — Providone-Iodine for periurethral preparation
  Arms: Betadine
Drug: Sterile water — Sterile water for periurethral preparation
  Arms: Sterile Water

SUMMARY:
The purpose of this study is to determine whether cleaning of the urethra, or external opening to the bladder, with sterile water (water that has been treated to remove bacteria and living organisms) vs Betadine also known as Povidone-Iodine (a medical grade cleaning solution) changes the rates of bacteria in the urine after a temporary catheter, or draining tube, is placed into the bladder. Chemical antiseptics, including Betadine, are the current standard of care. An additional goal of this study is to determine whether cleaning of the urethra, or external opening to the bladder, with sterile water vs betadine changes the amount of discomfort or pain patients experience with placement of a temporary catheter, or draining tube, in the bladder.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18+
* Patient undergoing in office straight catherization

Exclusion Criteria:

* History of culture proven recurrent urinary tract infection (2 in any 6-month period or 3 in any 12-month period)
* Urine Analysis with +Nitrites
* Catherization for any reason in the last 4 weeks
* History of Iodine allergy
* Patients unable to speak English
* Patient does not have the capacity to consent
* 2-3rd trimester pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2025-06-23 (Estimated); Primary Completion 2028-05-21 (Estimated); Study Completion 2028-05-21 (Estimated)

PRIMARY OUTCOMES:
Bacteruria | Within 2 weeks of the patients procedure date
  Bacteruria defined as the presence of bacteria within patient urine evaluated with urinalysis. Bacterial presence will be further characterized by colony forming unit count on urine culture.

SECONDARY OUTCOMES:
Urethral Pain | At the time of catherization
  Urethral pain at the time of catheterization rated by patients on a visual analog scale zero to ten with zero representing no pain and ten representing the worst pain of their life.

CONTACTS AND LOCATIONS:
Overall Officials: Ankita Gupta, MD, MPH, Principal Investigator — University of Louisville
Locations (2):
- United States (2):
  - UofL Physicians - Urogynecology Springs Urogynecology Office, Louisville, Kentucky
  - UofL Health - Urogynecology Mary & Elizabeth Hospital, Medical Plaza 4, Louisville, Kentucky

IPD SHARING:
Plan to Share IPD: No
Individual participant data collected in this study will be used solely for the purposes of completing this study

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-10): https://cdn.clinicaltrials.gov/large-docs/26/NCT07044726/Prot_SAP_000.pdf